CLINICAL TRIAL: NCT00680966
Title: Sequenced vs. Integrated Delivery of Treatment for Adolescent Depression and SUD
Acronym: Sequencing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA021357; 1R01DA021357 (NIH)
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Adolescent; Depression; Substance Use Disorders
Keywords: Treatment efficacy; Family therapy; Teens; Substance abuse; Substance dependence
MeSH Terms: conditions — Depression; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TX1 (Experimental): Functional Family Therapy (FFT) followed by Adolescent Coping With Depression (ACWD)
  Interventions: Behavioral: Adolescent Coping With Depression/Functional Family Therapy
- TX 2 (Experimental): ACWD (Adolescent Coping With Depression) followed by FFT (Functional Family Therapy)
  Interventions: Behavioral: Adolescent Coping With Depression/Functional Family Therapy
- TX 3 (Experimental): Combination of an augmented FFT and ACWD - Integrated treatment
  Interventions: Behavioral: Adolescent Coping With Depression/Functional Family Therapy

INTERVENTIONS:
Behavioral: Adolescent Coping With Depression/Functional Family Therapy — ACWD- Cognitive behavioral group therapy for depressed adolescents FFT - Family therapy to address substance use disorders in adolescents
  Other Names: FFT; ACWD

SUMMARY:
The purpose of this study is to determine whether it is more effective to treat adolescents, with diagnoses of both depression and substance use disorder, with a treatment addressing the substance use first and then treating the depression or to first treat the depression and then treat the substance use or whether treating both disorders simultaneously is most effective.

It is expected that treatment of both disorders at the same time will be the most effective.

DETAILED DESCRIPTION:
Comorbidity is a well established aspect of adolescent psychopathology. The majority of adolescents entering treatment have more than one condition. This study will evaluate service delivery methods of integrating empirically supported interventions for depression and non-nicotine substance use disorders (SUD)in an effort to improve treatment engagement, response, and maintenance of gains. The two examined interventions are the Adolescent Coping With Depression course (ACWD) and Functional Family Therapy (FFT).

This study will expand upon previous research by systematically treating both depression and SUD. Over a 5 year period, 180 adolescents with depression/SUD and their parents/guardians will be recruited in Oregon and New Mexico and randomly assigned to 1 of 3 conditions: (a) FFT followed by ACWD, (b) ACWD followed by FFT, or (c) an intervention combining and augmenting FFT and ACWD (Integrated Treatment). Each treatment arm will consist of 24 sessions provided over 20 weeks. Participants will be assessed at intake, after the provision of 6, 12 (Mid-treatment), 18 and 24 (Post-treatment)treatment sessions, and at 6 and 12 month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV-TR diagnosis of depression, defined as MDD, dysthymia, or substance-induced mood disorder meeting MDD or dysthymia symptom criteria
2. DSM-IV-TR diagnosis of one or more non-nicotine SUD
3. Some reported illicit drug use in the last 90 days
4. 13-17 years of age
5. parent or guardian willing to participate in study
6. basic English competency (ability to converse in English)

Exclusion Criteria:

1. Current and acute suicidal ideation at the level warranting inpatient treatment
2. current psychotic symptoms
3. the adolescent's sibling is already participating in the study
4. if on psychiatric medications, a significant change in dosage levels in the prior 4 weeks -

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2008-01; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Children's Depression Rating Scale | Intake, Mid-Treatment, Post, 6 months and 12 months follow-up

SECONDARY OUTCOMES:
Time Life Follow Back | Intake, Mid-Treatment, Post, 6 months and 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Rohde, Ph. D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States